CLINICAL TRIAL: NCT06266130
Title: A Randomized, Controlled, Two-arm Clinical Study to Evaluate Clinical Efficiency of 3MTM Digital Bonding Versus Direct Bonding
Brief Title: Digital Bonding vs. Direct Bonding Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum Orthodontics Corporation (Industry)
Responsible Party: Sponsor
Organization: Solventum US LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EM-11-050087
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Orthodontic Brackets

STUDY DESIGN:
Intervention Model Description: There are two groups, treatment group (digital bonding) and control group (direct bonding). Subjects will be enrolled and randomized into treatment or control group at each orthodontic practice.
Masking Description: Due to the nature of the devices, Investigator blinding is not feasible for the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment Group (Other): Digital Bonding Tray. Brackets will be bonded to each subject's teeth with a digital bonding tray.
  Interventions: Device: Treatment Group Digital Bonding Tray
- Control Group (Active Comparator): Direct bonding method. Brackets will be bonded to each subject's teeth by direct placement.
  Interventions: Device: Control Group Direct Bonding

INTERVENTIONS:
Device: Treatment Group Digital Bonding Tray — The Digital Bonding Tray is used in orthodontic treatment of misaligned teeth and provides a method to accurately position orthodontic brackets onto a patient's teeth simultaneously during a single procedure.
  Other Names: 3M Digital Bonding Tray
  Arms: Treatment Group
Device: Control Group Direct Bonding — The orthodontic brackets will be applied to Subject's teeth individually with direct bonding method.
  Other Names: Direct Bonding method
  Arms: Control Group

SUMMARY:
This is a prospective, 2-armed, randomized, multi-site clinical study to demonstrate that digital bonding is a more efficient treatment method than direct placement of brackets.

DETAILED DESCRIPTION:
Traditional Direct bonding bonds each bracket tooth by tooth individually. 3M digital bonding tray is a custom device which can have brackets pre-loaded according to the pre-determined placement by orthodontist prior to patient's arrival to the bonding appointment. This new bonding method allows orthodontist to bond an entire arch of brackets at once, significantly reducing chair time for patients. It is anticipated that patients in digital bonding group have shorter time spent for bonding brackets, less chair time, and fewer adjustment visits than those in direct bonding group.

The treatment arm utilizes a combination of the Digital Bonding Tray and pre adhesive-coated Brackets.

The study control arm will utilize the site's standard of care brackets (pre-adhesive-coated or non-coated) directly and individually applied to teeth. Roughly half of sites will utilize pre-coated brackets and the remaining sites will use uncoated brackets.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 12 years of age or older.
2. Subject is able and willing to provide their own informed Assent AND Subject or Legal Authorized Representative (LAR) is able and willing to sign the Informed Consent Form
3. Subject is able and willing to be available for all scheduled study visits.
4. The Subject is treatment-planned for required comprehensive orthodontic treatment for both arches using brackets.
5. Subject's current orthodontic treatment plan does not include extractions, orthognathic surgery, post-orthodontic restorative treatment (with the exception of minor spaces for tooth shaping post-orthodontic treatment), or temporary anchorage devices.
6. Subject has all permanent teeth erupted (dentition including second molars).
7. Subject has an Angle Class I or Class II (up to 3mm) molar and canine relationships.
8. The Subject has mild to moderate crowding (crowding less than 5 mm in each arch)
9. Subject has an overbite measuring between -1 mm (open bite) and 5 mm (deep bite).
10. The Subject's intra-oral scan must have been taken within 90 days of bracket placement.
11. The Subject is anticipated to complete treatment within 18 to 24 months.

Exclusion Criteria:

1. Subject has a history of adverse reaction to any materials used in this study.
2. Subject is pregnant or breast feeding.
3. Subject has advanced periodontal disease.
4. Subject has non-movable teeth (e.g., implants, bridges, ankylosed teeth).
5. Subject has more than 1 tooth excluded from the initial bonding (not including 2nd molars), e.g., no bracket placed on tooth due to position of the tooth at that point in time (tooth turned 90 degrees)
6. Subject will have more than 25% of the total number of brackets bonded to a non-enamel surface (e.g., restoration).
7. Subject has developmental abnormalities of the enamel (e.g., hypoplasia, moderate to severe fluorosis).
8. Subject has erupted 3rd molars.
9. Subject is, in the opinion of the investigator, unsuitable for enrollment in the study for reasons other than those specified in the above exclusion criteria.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Prep-and-bonding time | From the start of teeth preparation to the completion of bonding procedures.
  The duration (in minutes) for preparation of teeth, bracket positioning and bonding onto teeth

SECONDARY OUTCOMES:
Number of adjustment visits to complete treatment | Treatment duration from the completion of bonding visit to the bracket removal visit (18-24 months)
  Adjustment visits (visits with a bracket repositioning, arch wire compensation bend, and/or rebonding of a failed bracket).
Overall chair time | From initial bonding visit to the end of bracket removal visit.
  Sum of chair time for the initial application, necessary follow-up visits, and removal of treatment (in minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Lori Leitheiser, Study Chair — Solventum Orthodontics Corporation
Locations (5):
- United States (5):
  - The Orthodontic Studio, Glendale, California
  - Nadeau Orthodontics, Kennebunk, Maine
  - Northwell Health Physician Partners Dental Medicine at Great Neck, Great Neck, New York
  - Broadbent Orthodontics, Ogden, Utah
  - Larson Orthodontics, Altoona, Wisconsin

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD to other researchers.